CLINICAL TRIAL: NCT01897688
Title: A Phase 3 Single Center Study of Islet Transplantation in Non-uremic Diabetic Patients
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Daniel Borja-Cacho, Principal Investigator, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00059469
Record Dates: First submitted 2013-07-09; First posted 2013-07-12 (Estimated); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Type 1 Diabetes; Severe Hypoglycemic Unawareness
Keywords: Diabetes; Islet; Pancreas; Hypoglycemia; T1D; Transplant
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Hypoglycemia | interventions — Islets of Langerhans Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Islet Cell Transplant (Experimental): All qualified subjects will be put on United Network for Organ Sharing (UNOS) Islet Transplant wait list for potential islet cell transplant.
  Interventions: Biological: Islet Cell Transplant

INTERVENTIONS:
Biological: Islet Cell Transplant

SUMMARY:
Type 1 diabetes is an autoimmune disease in which the insulin-producing pancreatic beta cells are destroyed, resulting in poor blood sugar control. The purpose of this study is to determine the safety and effectiveness of islet transplantation, combined with immunosuppressive medications, specifically using Campath as induction, for treating type 1 diabetes in individuals experiencing hypoglycemia unawareness and severe hypoglycemic episodes.

DETAILED DESCRIPTION:
(T1D) Type 1 diabetes afflicts nearly 2 million people in the United States, most of them children or young adults. Untreated, it is a fatal disease. Exogenous insulin, administered by multiple injections or by a continuous subcutaneous (SC) infusion from a wearable pump, allow long term survival in those who develop the disease, and most who are treated in this way will have a very good health-related quality of life. However, insulin therapy does not provide normal glycemic control, and long term survivors commonly develop vascular complications such as diabetic retinopathy (the most common cause of adult blindness) and diabetic nephropathy (the most common indication for adult kidney transplantation). The Diabetes Control and Complications Trial (DCCT) established that these microvascular complications of diabetes can be prevented by maintaining near-normal glucose control in patients with T1D. However, this degree of control is not always achievable despite modern insulin analogs and delivery systems, and when achieved, it is invariably associated with episodes of insulin-induced hypoglycemia that can be life-threatening. A small minority of individuals with T1D develop hypoglycemia unawareness, a condition that is life-threatening, is associated with severe deterioration in quality of life and activity restriction, and is not amenable to medical therapy.

The hope of achieving near-normal glucose control without hypoglycemia in T1D has provided the impetus for developing effective strategies for β-cell replacement via pancreas or isolated islet transplantation. When successful, pancreas transplantation can normalize blood glucose(BG) in diabetic recipients, with associated stabilization and even reversal of microvascular complications. However, the risks of the procedure (an almost 10% early failure rate due to technical complications, anastomotic leak, bleeding, and infection) and the need for lifelong immunosuppression have in most centers limited the target population of this therapy to diabetics <50 years of age with minimal or no coronary artery disease, and at some centers pancreas transplant is offered only with concomitant kidney transplant. As a result, T1D patients in need of β-cell replacement are often excluded from whole pancreas transplantation. Islet transplantation, in contrast, is accomplished by a much simpler procedure in which the islets are infused into the portal vein. While this procedure is not without risk, the procedural morbidity is much less than that of whole pancreas transplantation.

On the other hand, whereas about 80% of whole pancreas transplant recipients will be insulin independent at one year after their transplant, <10% of 447 islet recipients transplanted between 1990 and 1999 achieved one year insulin independence. This was attributed to low engrafted islet mass combined with high metabolic demand imposed by glucocorticoids used to prevent rejection. In the year 2000, the group from Edmonton reported a series of 7 consecutive islet transplant recipients treated with islets from multiple donors and a glucocorticoid-free immunosuppressive regimen. These islet recipients were insulin free at follow-up ranging from 4.5 to 15 months. All of the recipients had experienced severe hypoglycemic episodes prior to transplant, and afterwards, none did. The efficacy of the Edmonton approach has now been confirmed by several other centers, and represents a major breakthrough in the field. However, it has also become clear that, in most islet recipients, there is loss of graft function over time; in Edmonton, insulin-independence rates have declined from 72% at one year to 28% by three years. A multicenter trial using the Edmonton protocol has both confirmed the results of the initial experience and raised questions relating to the expansion of the procedure to multiple centers, the toxicities of the immunosuppressive regimen, and the evaluation of the islet product.

In 2006, the NIH initiated several multi-center (Clinical Islet Transplantation Consortium) clinical trials of islet transplantation with the primary goal of establishing islet transplantation as a therapeutic treatment option for patients with type 1 diabetes either already have had a successful kidney transplant or with severe hypoglycemic events and good native renal function. The clinical protocol utilized for these trials improved from the Edmonton protocol in that it incorporates (1) T cell depletion anti-thymocyte antibody(16, 17); (2) peri-transplant anti-inflammatory therapy using Tumor Necrosis Factor (TNF)-a blockade; (3) aggressive control of glucose homeostasis after transplant with continuing, albeit reduced, insulin therapy; (4) short-term anticoagulation therapy peri-intraportal islet infusion. Northwestern is one of the clinical centers of the Consortium and has successfully transplanted a total of eighteen patients with twenty-six islet preparations using this protocol in the past two and half years.

The current study protocol modifies the protocol of the (CIT) Clinical Islet Transplantation consortium and substituted anti-thymocyte polyclonal antibody with alemtuzumab which has been shown to have efficacy in both pre-clinical model as well as clinical trials of allogeneic islet transplantation.

ELIGIBILITY:
Inclusion Criteria

1. Male and female patients age 18-65 years of age at consent
2. Ability to provide written informed consent
3. Mentally stable and able to comply with the procedures of the study protocol
4. Patients with T1D and insulin-dependent for at least 5 years fulfilling the following criteria:

   1. Absent stimulated c-peptide (<0.3 ng/mL) in response to a mixed meal tolerance test (MMTT; ensure 6 mL/kg body weight to a maximum of 360mL) measured at 60 and 90 min after the start of consumption
   2. Patients who have been followed by a qualified physician for diabetes management for a minimum of 12 months
   3. At least one episode of severe hypoglycemia in the past 12 months
   4. A Clarke score of 4 or more defining reduced awareness of hypoglycemia
5. Or, previous islet cell transplant recipients who have returned to partial or full insulin usage and are taking maintenance immunosuppression medications.

Exclusion Criteria

1. Body mass index (BMI) > 30
2. Insulin requirement of > 1.0 IU/kg/day
3. HbA1c > 10%
4. Calculated glomerular filtration rate (GFR) < 80mL/min for transplant-naïve patients (using subjects serum creatinine and the Chronic Kidney Disease Epidemiology Collaboration equation CKD-EPI) or 50mL/min for previously transplanted patients currently on immunosuppression
5. Macroalbuminuria >300 mg/g creatinine
6. Panel reactive anti-HLA antibodies> 50% by flow cytometry
7. For female subjects: positive pregnancy test, breast feeding or unwillingness to use effective contraceptive measures for the duration of the study.
8. Active infection including hepatitis B, hepatitis C, HIV, or tuberculosis (TB)
9. Negative Epstein-Barr Virus (EBV) by IgG
10. Any history of malignancy except resected squamous or basal cell carcinoma
11. Alcohol or substance abuse
12. Baseline Hb below the lower limit of normal
13. International normalized ratio >1.5 and long term anticoagulant therapy
14. Clinically significant coronary artery disease
15. Elevated liver function tests >1.5 times upper limit of normal
16. Symptomatic cholecystolithiasis
17. Gastrointestinal disorders interfering with ability to absorb oral medications
18. Uncontrolled hyperlipidemia (LDL cholesterol >130 mg/dL and/or triglycerides >200 mg/dL)
19. Chronic corticosteroid use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-06; Primary Completion 2025-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
To demonstrate the safety and efficacy of islet transplantation under alemtuzumab induction for treatment of Type-1 Diabetes (T1D) in subjects with hypoglycemia unawareness and a history of severe hypoglycemic episodes. | Two years after the final islet transplant.
  To assess the efficacy of islet cell transplantation under alemtuzumab induction immunosuppression on the proportion of subjects with a change in HbA1c and free of severe hypoglycemic events through two years after the final islet transplant.

SECONDARY OUTCOMES:
To relate clinical transplant outcomes based upon islet quantity/quality to organ donor characteristics | Two years after the final islet transplant.
  To assess the proportion of insulin-independent subjects at two years after the final islet transplant.
To relate clinical transplant outcomes based upon islet quantity/quality to organ donor characteristics. | Two years after the final islet transplant.
  To compare islet graft outcome between alemtuzumab induction and historical anti-thymocyte induction groups.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Borja-Cacho, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States